CLINICAL TRIAL: NCT01744600
Title: Music Therapy in Methodist Homes: a Cluster Randomised Controlled Trial Including Mixed Methods Analysis Investigating the Efficacy of the Impact of a Music Therapy Programme on Caring for People With Dementia Who Have Behavioural Symptoms.
Brief Title: Music Therapy in Methodist Homes: a Study Investigating the Impact of a Music Therapy Programme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Methodist Homes for the Aged (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MTRP-301013
Record Dates: First submitted 2012-11-30; First posted 2012-12-06 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Dementia
Keywords: Dementia; Music Therapy
MeSH Terms: conditions — Dementia | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music Therapy (Experimental): Participants in the experimental group will receive one active individual music therapy session each week for 22 weeks. Each session will last thirty minutes.
  Interventions: Behavioral: Music Therapy
- Control (No Intervention): Participants in the control group will receive normal, standard daily care for the 22 week period.

INTERVENTIONS:
Behavioral: Music Therapy — The music therapy intervention will consist of individual active music therapy session each week for a period of 22 weeks. Each session will last 30 minutes.
  Arms: Music Therapy

SUMMARY:
The study is a cluster randomised control trial, which aims to investigate the effectiveness of music therapy in minimising Behavioural and Psychological Symptoms of Dementia (BPSD) in older adults with dementia. In particular, the study aims to identify the main components of music therapy that are key in achieving this. The study will also explore carers' perceptions of music therapy, and investigate whether carers become more attentive to patients' needs and more able to manage patients' BPSD as a result of the music therapy programme.

DETAILED DESCRIPTION:
While music therapy has been noted to be an effective intervention in decreasing agitation and disruptive behaviour in adults with dementia (Livingston et al, 2005), these effects have only been demonstrated during and immediately after sessions, arguably due to the progressive nature of dementia. To achieve long-lasting therapeutic change, it seems necessary to consider the specific elements that work in music therapy, and extract them for use within other activities. It is hypothesised that the use of such elements within additional activities and care provision, alongside regular music therapy sessions, may result in decreasing residents' BPSD for a longer duration of time.

Little research has been carried out that specifically identifies the key elements of music therapy which contribute to its efficacy within the field of dementia. This study aims to support existing evidence highlighting the significance of using music therapy within dementia care, and, importantly, identify what elements are principally involved in producing changes in behaviour and levels of well-being. The study will also incorporate the collection of dementia residents' physiological data, specifically their Electrodermal Activity (EDA), during therapy sessions. This will be measured by recording participants' levels of skin conductance (microSiemens/cm); this is controlled by the Sympathetic Nervous System and roughly thought of as the Fight or Flight system. Many efforts have been made to explore how skin conductance indicates the levels of emotional arousal, for example, high skin conductance indicates excitement or stress; low skin conductance indicates sadness or calmness. (Poh et. al., 2010; 2012; Van Dooren et. al., 2012). The skin conductance data is proposed to help identify the key elements and observable phenomena of the videoed music therapy sessions showing reduced presentation of BPSD.

If the current study is able to identify such elements, these findings will enable future research to investigate more comprehensively how these can be transplanted into other activities to optimise their effects.

Participants will be recruited from two residential Methodist Homes, and using a cluster randomized control design, will be allocated to either the control group on intervention group. Participants in the control group will receive standard daily care for 22 weeks. Participants in the intervention group will, in addition to daily standard care, receive one session of individualised active music therapy once a week for a period of 22 weeks.

Music therapy sessions will last 30 minutes. During the session the participant will wear a 'Q-sensor' device around their wrist, which will record their skin conductance levels. Each session will be video-recorded.

A communication system will be employed after each therapy session, in which video clips of the session demonstrating the participant engaging in an interaction or expression will be presented to care staff. This process will aim to demonstrate to staff how Behavioural and Psychological Symptoms of Dementia (BPSD) are minimised by music therapy techniques, the possible causes of BPSD, and how the therapist has made use of the participants' remaining abilities to enhance and facilitate their involvement and interpersonal communication within sessions.

The primary outcome measure will be the Neuropsychiatric Inventory, a standardised questionnaire used to assess the psychopathology of dementia patients. This will be carried out with residents' keyworkers at the following time points: as a baseline measure in the 2 weeks prior to the commencement of the music therapy intervention period, then at weeks 11-12, weeks 21-22 and as a follow-up at weeks 27-28. There will be three secondary outcome measures:

1. dementia care mapping, an observational tool used to assess the quality of care delivered by staff. This will be carried out at baseline in the 2 weeks prior to the commencement of the music therapy intervention; then at weeks 11-12; weeks 21-22; and as a follow-up at weeks 27-28.
2. microanalysis of video recordings of music therapy sessions, in conjunction with data on participants' arousal levels during sessions, measured by a skin conductance device worn on the wrist. This will take place each week after each music therapy session for the duration of the 22 week intervention period.
3. grounded-theory based interviews. These will be carried out with care staff during weeks 23 and 25 to explore carers' perceptions of music therapy.

Further analysis of video recordings of sessions will be conducted following the completion of the 22-week period of music therapy treatment to further investigate key moments within sessions.

ELIGIBILITY:
31 participants are proposed to be recruited in total. This number comprises 16 resident participants, 14 staff participants and 1 music therapist.

The music therapist has already been recruited for the study and works within for the organisation's music therapy service in the two homes to be used as the research sites. The inclusion and exclusion criteria for staff and residents are outlined below.

Inclusion Criteria:

The proposed inclusion criteria for care home residents are as follows:

* Participants will be a resident at one of the two residential homes identified as the research sites, in one of the two house units that will be used in the project in each home.
* Participants will have a diagnosis of dementia
* Participants will display at least one symptom of BPSD
* Participants will be at least 40 years of age

The proposed inclusion criteria for staff participants are as follows:

* Staff participants will have at least three months' experience of working with the resident participant(s)
* Staff participants will have an in-depth knowledge of the resident participant(s) in a 'keyworker' role

Exclusion Criteria:

The proposed exclusion criterion for care home residents is as follows:

• Residents will be excluded if their health appears to be at a risk which raises concerns regarding their sustained involvement within the study, apparent from a general health examination with their General Practitioner

The proposed exclusion criteria for care staff participants is as follows:

* Staff who have not worked with the resident participant(s) in a 'keyworker' role for at least three months.
* Staff who would be unable to regularly work on the specific days they would be required within the home.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Neuropsychiatric Inventory | At baseline in the 2 weeks prior to the music therapy intervention, then at weeks 11-12, weeks 21-22 and as a follow-up at week 27-28.
  The NPI assesses the neuropsychiatric symptoms and pathology of patients with Alzheimer's disease and other neurodegenerative disorders.
  Ten behavioural areas (delusions, hallucinations, agitation/aggressions, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability and aberrant motor behaviour) and two neuro-vegetative areas (sleep and night-time behaviour disorders, and appetite and eating disorders) are assessed.
  Changes in these areas of behaviour over the two weeks prior to interview will be investigated. This project will employ the version of the NPI which has been developed for use within institutional settings (NPI-NH). The interviews will be conducted with an informed professional caregiver.

SECONDARY OUTCOMES:
Dementia Care Mapping | At baseline in the 2 weeks prior to the start of the music therapy intervention, then at weeks 11-12, weeks 21-22 and as a follow-up at weeks 27-28.
  Dementia Care Mapping (DCM) is an observational tool used within institutional settings that aims to provide information on residents' well-being and the quality of care delivered by staff. During a mapping session, the mapper(s) record resident's behaviours, mood, engagement and interactions with staff over a defined time period, within a communal area. For the purposes of this study, participants will be observed for two consecutive hours beginning from one hour prior to lunch.
  Each construct of behaviour, mood and engagement is systematically coded within 5-minute time frames, and the resulting data set is then analysed to give an overall 'wellbeing' level. Staff-resident interactions are recorded as and when they occur, according to type and potential for well-being, and are named as 'personal detractors' or 'personal enhancers'. These aim to give an overall picture of the level and quality of person-centred-care being delivered.
Grounded theory-based interviews | The two sets of interviews will be carried out during weeks 23 and 25.
  Two sets of Grounded Theory-based interviews will be carried out with care staff to explore their perceptions of music therapy. Grounded theory, developed by Glaser and Strauss (1967), is an inductive methodology by which theories are systematically generated from data without the use of pre-determined hypotheses. The process consists of a period of data collection; 'coding', in which themes and categories within the data are identified; 'memo-ing', the writing up of theoretical ideas on the codes and their relationships; and 'sorting' the memo's into an outline of the emerging theory. The phases of data collection, coding and memo-ing are ongoing and overlap, enabling an organic, flexible approach for themes to emerge within.
Microanalysis of video recordings of sessions | Video recordings of music therapy sessions will be analysed for the duration of the 22 week intervention period, immediately after each weekly music therapy session.
  The method of microanalysis employed in this project will follow a similar procedure to those outlined by Ridder (2003), De Backer, (2005) and Trondalen (2005).
  After each music therapy session, the research assistant and music therapist will play back the video recording and transcribe the interactions and expressions of the therapist and client. An Excel file developed by the Lead Researcher for this purpose will be used during this process.
  The session will be divided into one-second timeframes and data will be recorded separately for both the therapist and client. For each timeframe that an expression is observed, a code will be chosen and inputted according to the nature of the client or therapist's expressions: musical, verbal, non-verbal or mixed. 'Special events' will also be recorded as and when they happen; these are sudden behaviours or changes in behaviours that raise questions and reflect something significant about the experience of the client in that moment.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hung Hsu, MA, Principal Investigator — Methodist Homes
Locations (2):
- United Kingdom (2):
  - The Homestead, Carterton, Oxfordshire
  - Fitzwarren House, Swindon

REFERENCES:
- [Background] Livingston G, Johnston K, Katona C, Paton J, Lyketsos CG; Old Age Task Force of the World Federation of Biological Psychiatry. Systematic review of psychological approaches to the management of neuropsychiatric symptoms of dementia. Am J Psychiatry. 2005 Nov;162(11):1996-2021. doi: 10.1176/appi.ajp.162.11.1996. PMID 16263837
- [Background] Fossey J, Lee L, Ballard C. Dementia Care Mapping as a research tool for measuring quality of life in care settings: psychometric properties. Int J Geriatr Psychiatry. 2002 Nov;17(11):1064-70. doi: 10.1002/gps.708. PMID 12404656
- [Background] Poh MZ, Swenson NC, Picard RW. A wearable sensor for unobtrusive, long-term assessment of electrodermal activity. IEEE Trans Biomed Eng. 2010 May;57(5):1243-52. doi: 10.1109/TBME.2009.2038487. Epub 2010 Feb 17. PMID 20172811
- [Background] Poh MZ, Loddenkemper T, Reinsberger C, Swenson NC, Goyal S, Sabtala MC, Madsen JR, Picard RW. Convulsive seizure detection using a wrist-worn electrodermal activity and accelerometry biosensor. Epilepsia. 2012 May;53(5):e93-7. doi: 10.1111/j.1528-1167.2012.03444.x. Epub 2012 Mar 20. PMID 22432935
- [Background] van Dooren M, de Vries JJ, Janssen JH. Emotional sweating across the body: comparing 16 different skin conductance measurement locations. Physiol Behav. 2012 May 15;106(2):298-304. doi: 10.1016/j.physbeh.2012.01.020. Epub 2012 Feb 4. PMID 22330325
- [Background] Glaser, B. G. and Strauss, A. L., 1967. The discovery of grounded theory: strategies for qualitative research. Chicago: Aldine.
- [Background] De Backer, J., 2005. The transition from sensorial impression to a musical form ( proto-symbolism) in psychotic patients in a music therapeutic process. Ph. D. Aalborg University.
- [Background] Ridder, H.M.O., 2003. Singing dialogue: Music therapy with persons in advanced stages of dementia. A case study research design. Ph. D. Aalborg University.
- [Background] Trondalen, G., 2005. Significant moments" in music therapy with young persons suffering from anorexia nervosa. Music Therapy Today, 6, pp. 396-429.
- [Derived] Hsu MH, Flowerdew R, Parker M, Fachner J, Odell-Miller H. Individual music therapy for managing neuropsychiatric symptoms for people with dementia and their carers: a cluster randomised controlled feasibility study. BMC Geriatr. 2015 Jul 18;15:84. doi: 10.1186/s12877-015-0082-4. PMID 26183582